CLINICAL TRIAL: NCT04722575
Title: "NEOadjuvant Plus Adjuvant Therapy With Combination or Sequence of Vemurafenib, cobImetinib, and atezolizuMab in Patients With High-risk, Surgically Resectable BRAF Mutated and Wild-type Melanoma"
Brief Title: Combination or Sequence of Vemurafenib, Cobimetinib, and Atezolizumab in High-risk, Resectable Melanoma
Acronym: NEO-TIM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Melanoma Onlus (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEO-TIM
Record Dates: First submitted 2021-01-18; First posted 2021-01-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Melanoma
Keywords: resectable melanoma; BRAF mutated; high risk melanoma; wild type
MeSH Terms: conditions — Melanoma | interventions — cobimetinib; Tablets; Vemurafenib; atezolizumab; Injections

STUDY DESIGN:
Intervention Model Description: The study will be conducted according to an open-label, randomized, not comparative phase II design. Three arms for a total of 88 patients will be considered.
  BRAF mutated patients will be randomized in two arms: Arm A and Arm B (27 patients per arm). BRAF WT patients will be included in Arm C (34 patients).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ARM A (Experimental): Arm A BRAF mutated patients. Over a period of 6 weeks (1) + (2):
  1. Vemurafenib 960 mg bid p.o. from week 1 to week 6.
  2. Cobimetinib 60 mg qd p.o. from week 1 to week 3 and week 5 to week 6. Week 4 off.
  After surgery and a second screening period (up to six weeks): Atezolizumab 1200 mg IV for 52 weeks
  Interventions: Drug: Cobimetinib 20 MG Oral Tablet; Drug: Vemurafenib 240 Mg Oral Capsule; Drug: Atezolizumab 1200 MG in 20 ML Injection
- ARM B (Experimental): Arm B BRAF mutated patients. Over a period of 6 weeks (1) + (2) + (3):
  1. Vemurafenib 720 mg bid p.o. from week 1 to week 6.
  2. Cobimetinib 60 mg qd p.o. from week 1 to week 3 and from week 5 to week 6. Week 4 off.
  3. Atezolizumab 840 mg IV for 2 cycles (day 1 of week 4 and day 1 of week 7).
  After surgery and a second screening period (up to six weeks): Atezolizumab 1200 mg IV for 52 weeks
  Interventions: Drug: Cobimetinib 20 MG Oral Tablet; Drug: Vemurafenib 240 Mg Oral Capsule; Drug: Atezolizumab 1200 MG in 20 ML Injection
- ARM C (Experimental): Arm C BRAF WT patients. Over a period of six weeks (1) + (2):
  1. Cobimetinib 60 mg qd p.o. from week 1 to week 3 and from week 5 to week 6,
  2. Atezolizumab 840 mg IV for 2 cycles (day 1 of week 1 and day 1 of week 4).
  After surgery and a second screening period (up to six weeks): Atezolizumab 1200 mg IV for 52 weeks
  Interventions: Drug: Cobimetinib 20 MG Oral Tablet; Drug: Atezolizumab 1200 MG in 20 ML Injection

INTERVENTIONS:
Drug: Cobimetinib 20 MG Oral Tablet — Cobimetinib 60 mg qd p.o. from week 1 to week 3 and week 5 to week 6. Week 4 off.
  Other Names: Cotellic
Drug: Vemurafenib 240 Mg Oral Capsule — 960 (arm A) /720 (arm B) mg bid p.o. from week 1 to week 6.
  Other Names: Zelboraf
  Arms: ARM A; ARM B
Drug: Atezolizumab 1200 MG in 20 ML Injection — 840 mg IV for 2 cycles for Arm B and C. After surgery in all arms 1200 mg IV for 52 weeks
  Other Names: Tecentriq

SUMMARY:
Neoadjuvant plus adjuvant treatment with target therapy and immunotherapy given in combination or sequence may have an anti-tumour activity and may reduce the risk of relapse in patients with high-risk resectable melanoma (stage III B / C / D and oligometastatic stage IV).

DETAILED DESCRIPTION:
Melanoma represents a considerable health burden and an ongoing area of unmet need in oncology. Despite melanoma accounts for only 1% of diagnosed skin cancers, it is the cause of most skin cancer-related deaths. Until recently, limited effective treatment options were available to patients with advanced melanoma. Historically, response rates to conventional chemotherapy and immunomodulation therapy (interleukin-2 or interferon-γ) have been reported at approximately 5-19%.

Adjuvant immune checkpoint blockade (ICB) and target therapy improve outcomes of patients with high-risk resectable melanoma. It has recently been demonstrated that treatment with neoadjuvant and adjuvant targeted therapy (dabrafenib and trametinib) is associated with a high pathologic complete response (pCR) rate and improved outcomes over surgery alone. However, treatment with ICB has not been well studied in the neoadjuvant setting, despite preclinical studies suggesting that neoadjuvant administration of ICB is associated with improved survival and enhanced anti-tumour immune responses compared to the same therapy administered in the adjuvant setting.

The advantage of neoadjuvant trials is the availability of blood and tumour tissue samples before and after systemic therapy for the conduct of novel mechanistic and biomarker studies in the circulation and the tumour microenvironment.

Prospective neoadjuvant clinical trials with targeted (dabrafenib/trametinib combo) or immunotherapeutic agents (nivolumab alone or nivolumab/ipilimumab combo) and combinations are now running in a subgroup of highrisk melanoma patients with pooled overall promising preliminary results of high rates of pathologic complete responses (pCRs, 30-50%) and early data of positive correlation between pCR and relapse-free survival. Based on the available results to date, we aim to conduct a randomized, noncomparative phase II trial to define the role of neoadjuvant plus adjuvant target and immunotherapy, given in combination or sequence, in patients with high risk surgically resectable melanoma.This approach has the potential to define whether neoadjuvant treatment has antitumour activity and whether it reduces the risk of relapse after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged ≥18 years;
2. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form;
3. Patients must have histologically or cytologically confirmed Stage IIIB/C/D or oligometastatic stage IV1 resectable melanoma. The definition of resectability can be determined by the patient's surgical oncologist and verified via discussion at Multidisciplinary Tumour Conference attended by melanoma medical and surgical oncology staff. Resectable tumours are defined as having no significant vascular, neural or bony involvement. Only cases where a complete surgical resection with tumour-free margins can safely be achieved are defined as resectable;
4. All patients must have a BRAF V600E/K mutation status known;
5. Patients must be medically fit enough to undergo surgery as determined by the surgical oncology team;
6. Patients must have measurable disease, defined by RECIST 1.1;
7. ECOG performance status 0-1; *
8. Patients must have organ and marrow function
9. Absence of any psychological, familiar or social condition that may affect compliance with study protocol and schedule follow-up;
10. Female subjects of childbearing potential must have a negative pregnancy test result at baseline and must practice a reliable method of contraception for the total study duration plus 23 weeks (i.e. 30 days plus the time required for experimental drugs to undergo five half-lives) after the last dose of experimental drugs; *
11. Men who are sexually active with women of childbearing potential must practice a reliable method of contraception for the total study duration plus 31 weeks (i.e. 80 days plus the time required for experimental drugs to undergo five half-lives) after the last dose of experimental drugs.

Exclusion Criteria:

1. Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug; *
2. Prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, thyroid cancer (except anaplastic) or any cancer from which the patient has been disease-free for 2 years;
3. Any major surgery within the last 3 weeks;
4. Pregnancy and/or breast feeding or of childbearing potential and not practicing a reliable method of birth control;*
5. Unwillingness or inability to follow the procedures required in the protocol; *
6. Uncontrolled diabetes, hypertension or other medical conditions that may interfere with assessment of toxicity;*
7. Current use of anticoagulants (warfarin, heparin, direct thrombin inhibitors) at therapeutic levels*
8. Patients with a history of uncontrolled cardiovascular or interstitial lung disease and evidence or risk of retinal vein occlusion or central serous retinopathy;
9. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of treatment; *
10. Prior BRAF or MEK directed therapy; patients who have received prior interferon are eligible;
11. History of retinopathy or any finding at ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy, retinal vein occlusion (RVO), or neovascular macular de generation;
12. Presence of any of the following risk factors for RVO: a) Uncontrolled glaucoma with intraocular pressures ≥ 21mmHg; b) Serum cholesterol ≥Grade 2; c) Hypertriglyceridemia ≥ Grade 2; d) Hyperglycaemia (fasting) ≥Grade 2;
13. Correct QT interval > 450msec to baseline, history of congenital long QT syndrome;
14. Uncontrolled medical condition among which endocrine disorders (such as hypothyroidism, hyperthyroidism and diabetes mellitus);
15. Other severe medical or psychiatric conditions (like depression) or abnormalities of laboratory tests that may increase the risk associated with study participation or the assumption of Vemurafenib, Atezolizumab and Cobimetinib or that may interfere with the interpretation of study results, which in the judgment of the Investigator can make the patient not eligible for the study;
16. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, cerebrovascular accident or transient ischemic attack, pulmonary embolism, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent;
17. History of active primary immunodeficiency;
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of IMP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IMP and up to 30 days after the last dose of IMP; *
19. Prior treatment with an anti- PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody;
20. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients;
21. Positive test for HBV sAg or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection;
22. Known history of testing positive for HIV or known AIDS;
23. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) rate (Centrally/Independently determined) | At surgery (from week 8 to week 9)
  Defined as the lack of all signs of cancer in tissue samples removed during surgery

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | At 2-years, 3-years and at the end of the study
  Defined as the time from randomisation to recurrence event or last follow-up
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  Defined as the time from the date of randomisation to the date of death due to any cause
pORR | At surgery (from week 8 to week 9) after neoadjuvant treatment and at disease relapse up to 5 years
  Defined as the sum of pathologic complete responses (pCRs), near pathologic complete responses near pCRs) and pathologic partial responses (pPRs).
Safety - adverse events | Continuosly during the trial while on treatment or within 30 days after the last study treatment
  All AEs, Grade 3 to 4 AEs, serious adverse events (SAEs), deaths, AEs of special interest (AESIs), and AEs leading to treatment discontinuation or withdrawal from the study
Molecular and immunophenotypic changes | At baseline, prior to surgery, every 12 weeks during adjuvant treatment and at the disease relapse up to 5 years
  Immunoscore, Circulating cytokines and chemokines profiling, Metabolomic profiling,Tumour mutational burden, Myeloid-derived suppressors cells, immune cell subtypes expression and lymphocyte activation, Additional analysis of protein levels (i.e. CCR5), DNA mutations, and/or mRNA analysis

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Ascierto, Study Chair — Fondazione Melanoma Onlus
Locations (6):
- Italy (6):
  - Ospedale S.M. Annunziata - Azienda USL Toscana Centro, Bagno a Ripoli, Firenze
  - IRCCS - Istituto Scientifico Romagnolo per la Cura e lo Studio dei Tumori (I.R.S.T) S.r.l., Meldola, Forlì-Cesena
  - Fondazione I.R.C.C.S. Istituto Nazionale dei Tumori, Milan, Milano
  - Istituto Nazionale per lo Studio e la Cura dei Tumori "Fondazione Giovanni Pascale", Naples, Naples
  - Istituto Oncologico Veneto, Padua, Padova
  - IRCCS San Martino - IST, Genova

IPD SHARING:
Plan to Share IPD: No